CLINICAL TRIAL: NCT05524532
Title: Effect of Immulina Supplements on Inflammatory Biomarkers Correlated With Clinical Symptoms in Patients With Long COVID (PASC)
Brief Title: Effects of Immulina TM Supplements With PASC Patients
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Mississippi Medical Center (Other)
Collaborators: National Institute of General Medical Sciences (NIGMS) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: 2022-272; U54GM115428 (NIH)
Record Dates: First submitted 2022-07-18; First posted 2022-09-01 (Actual); Last update posted 2025-08-14 (Actual); Status verified 2025-08

CONDITIONS: Post Acute COVID-19 Syndrome
Keywords: Immulina; Post Acute Covid-19 Syndrome; Inflammation; Natural Dietary Supplement
MeSH Terms: conditions — Post-Acute COVID-19 Syndrome; Inflammation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Immulina TM 800 mg/day (Experimental): Immulina Dietary supplementation (200 mg per capsule) 2-200 mg capsules given by mouth in the morning and 2-200 mg capsules given by mouth in the evening for 8 weeks duration
  Interventions: Drug: Immulina TM
- Placebo (Placebo Comparator): inert capsules; 2 capsules given by mouth in the morning and 2 capsules given by mouth in the evening for 8 weeks duration
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Drug: Immulina TM — Immulina TM is a highly standardized extract derived from various preparations of Spirulina, a cyanobacterium, marketed as a dietary supplement and has been utilized in several clinical studies describing its immunopotentiiating properties.
  Other Names: Spirulina
  Arms: Immulina TM 800 mg/day
Dietary Supplement: Placebo — Placebo is an inert form of cellulose acetate.
  Arms: Placebo

SUMMARY:
This is a multi-site study that will try to determine the effects of Immulina ™, a natural dietary supplement, on blood chemicals associated with inflammation that are often increased in patients with long COVID (also called PASC).

DETAILED DESCRIPTION:
This is a randomized, double-blind placebo controlled pilot study designed to determine effect size on altering blood inflammatory biomarkers and anti SARS-CoV-2-specific adaptive response including memory T cell, memory B cells and antiviral antibody titers. The participants will have a variety of clinical manifestations that will include varying degrees of fatigue, cognitive dysfunction and other PASC-related symptoms. Individuals will be randomized by site to receive either Immulina or placebo given daily for 8 weeks followed by a 4 week observation off supplement.

ELIGIBILITY:
Inclusion Criteria:

* Males and females, 18 to 99 years old
* If female of child bearing potential, using acceptable means of birth control or postmenopausal for at least two years
* Body temperature between 36.1°C and 37.7°C.
* Has completed the 4-week washout period (if applicable), i.e., has refrained from using internally-consumed dietary supplements prior to Study Day 1 and through the completion of the study
* A minimum of 2 hours fasting (except water) prior to all of the blood draws
* Willing and able (in the opinion of study staff) to comply with all study requirements, including swallowing size 4 capsules (approximately 0.5" long and 0.25" diameter) and having phlebotomy
* Good written and verbal English skills; able to follow instructions (in the investigator's opinion)
* Not participating in a clinical study, currently or within the last 30 days
* Signed informed consent

Exclusion Criteria:

* Pregnant or lactating
* Digestive tract disorders or conditions, such as (but are not limited to): ulcers, ulcerative colitis, Crohn's disease, gastric bypass, colostomy, ischemic colitis, gastroesophageal reflux disease (GERD), irritable bowel disease (IBD), diverticulitis that would be expected to impact on the oral disposition of the Immulina dietary supplement
* Existence of any surgical and/or medical condition, significant disease or disorder, or any finding that may, in the judgment of the investigator, put the volunteer at risk or compromise study participation.
* Any blood-thinning or clotting concomitant medication (prescription anticoagulants)
* Donation or loss of 400 mL or more of blood within 8 weeks of Study Day 1 or unwilling to abstain from donation of blood during the study
* Known or suspected allergy or sensitivity to Immulina, cellulose
* History of drug or alcohol abuse within the last 12 months

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 101 (Actual)
Dates: Start 2023-07-20 (Actual); Primary Completion 2025-07-29 (Actual); Study Completion 2025-07-29 (Actual)

PRIMARY OUTCOMES:
Plasma IL-6 (Interleukin 6, pg/mL) | 12 weeks
  Differences in Interleukin 6 from baseline to 12 weeks
Plasma CRP (C-Reactive Protein, ng/mL) | 12 weeks
  Differences in C-Reactive Protein from baseline to 12 weeks.
Plasma D-Dimer, pg/mL | 12 weeks
  Differences in D-Dimer from baseline to 12 weeks.

SECONDARY OUTCOMES:
PROMIS-29 | 12 weeks
  Differences in questionnaire PROMIS-29, Domain T-scores PROMIS-29 is a collection of short forms containing a fixed number of items from the same 7 PROMIS domains (physical function, anxiety, depression, fatigue, sleep disturbance, ability to participate in social roles and activities, and pain interference) plus a single item on pain intensity. They assess all domains over the past seven days except the Physical Function, which has no timeframe specified. Four questions asked for each of 7 domains, plus the single pain intensity item and scored separately, yielding a total of 7 domain scores. The final score is represented by the T-Score, a standardized score with a mean of 50 and a standard deviation [SD] of 10. High scores mean more of the concept being measured (e.g., more fatigue, more Physical Function).
FSS | 12 weeks
  Differences in Fatigue Severity Scale (FSS) questionnaire between baseline to 12 weeks
  Changes in questionnaire FSS, units on a scale, results that reflect PASC-associated symptoms of fatigue, neurocognitive dysfunction, dyspnea and/or other symptoms.
  The questionnaire FSS contains nine statements that rate the severity of fatigue symptoms. Respondents rate their fatigue severity during the past seven days using a 7 point rating scale. A low value (e.g.1) indicates strong disagreement with the statement, whereas a high value (e.g.7) indicates strong agreement. A total score of less than 36 suggests that the respondent may not be suffering from fatigue. A total score of 36 or more suggests that the respondent may need further evaluation by a physician.
SBQ-LC TM | 12 weeks
  Differences in The Symptom Burden Questionnaire for Long COVID (SBQ-LC TM) questionnaire between baseline to 12 weeks
  Changes in questionnaire SBQ-LC TM (units on a scale) results that reflect PASC-associated symptoms of fatigue, neurocognitive dysfunction, dyspnea and/or other symptoms .
  SBQ-LC TM (version 1.0) is a modular instrument measuring patient reported outcomes and is composed of 17 independent scales with promising psychometric properties. Respondents rate their symptom burden during the past seven days using a dichotomous response or 4 point rating scale. Each scale provides coverage of a different symptom domain and returns a summed raw score that can be transformed to a linear (0-100) score. Higher scores represent higher symptom burden.
SARS-CoV-2-specific antibody responses | 12 weeks
  Differences in SARS-CoV-2-specific antibody immune responses: Receptor Binding domain (RBD) and Nucleocapsid (NP) antibody responses between baseline and 12 weeks
SARS-CoV-2-specific immune responses on memory T cell levels | 12 weeks
  Differences in SARS-CoV-2-specific immune responses on memory T cell levels between baseline and 12 weeks
SARS-CoV-2-specific immune responses on memory B cell levels | 12 weeks
  Differences in SARS-CoV-2-specific immune responses on memory B cell levels between baseline and 12 weeks
Natural Killer cell (NK)-mediated cytotoxicity | 12 weeks
  NK cell-mediated cytotoxicity is characterized by cytolysis of a CSFE-labeled (K562) by effector cells (NK cells). Labeled K562 are cultured with NK cells for a period of time, then all cells labeled with a live-dead stain, 7-AAD. The cytolytic actively is expressed as the percent dead K562.
  Difference in cytolytic activity (%dead K562) from baseline to 20 weeks.
Natural Killer (NK) cell count | 12 weeks
  Difference in NK cell counts from baseline to 20 weeks.
Cytolytic T lymphocyte (CTL) number | 12 weeks
  Difference in CTL cell number from baseline to 20 weeks.
serum Interferon alpha, pg/mL | 12 weeks
  Difference in Interferon alpha from baseline to 20 weeks.
serum Interferon gamma, pg/mL | 12 weeks
  Difference in Interferon gamma from baseline to 20 weeks.

CONTACTS AND LOCATIONS:
Overall Officials: Gailen D Marshall, Jr., MD, PhD, Principal Investigator — University of Mississippi Medical Center
Locations (9):
- United States (8):
  - University of Hawaii, Honolulu, Hawaii
  - Pennington Biomedical Research Center, Baton Rouge, Louisiana
  - Louisiana State University, New Orleans, Louisiana
  - MaineHealth, Portland, Maine
  - University of Mississippi Medical Center, Jackson, Mississippi
  - University of Nebraska Medical Center, Omaha, Nebraska
  - University of Oklahoma, Oklahoma City, Oklahoma
  - West Virginia University, Morgantown, Virginia
- University of Puerto Rico, San Juan, Puerto Rico, Puerto Rico

IPD SHARING:
Plan to Share IPD: No